CLINICAL TRIAL: NCT02336581
Title: Effectiveness of Psychosocial Treatment for Inpatients With Psychosis
Brief Title: Researching the Effectiveness of Acceptance-Based Coping During Hospitalization
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Brandon Gaudiano, Research Psychologist/Associate Professor, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1411-001; 5R34MH097987-02 (NIH)
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Psychosis; Schizophrenia
Keywords: Acceptance and Commitment Therapy; Mindfulness; Inpatients; Psychiatric Hospitalization
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acceptance and Commitment Therapy (ACT) (Experimental): ACT which includes individual and group sessions during hospitalization and follow-up phone contacts the first month following hospital discharge.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Enhanced Treatment as Usual (eTAU) (Active Comparator): Enhanced treatment as usual (eTAU) which includes other individual and group sessions during hospitalization and follow-up phone contacts the first month following hospital discharge.
  Interventions: Behavioral: Enhanced Treatment as Usual (eTAU)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — individual + group + follow-up phone contacts
  Arms: Acceptance and Commitment Therapy (ACT)
Behavioral: Enhanced Treatment as Usual (eTAU) — individual + group + follow-up phone contacts
  Arms: Enhanced Treatment as Usual (eTAU)

SUMMARY:
To test the effectiveness of Acceptance and Commitment Therapy (ACT) versus enhanced Treatment as Usual (eTAU) delivered by hospital staff for inpatients with psychotic-spectrum disorders.

DETAILED DESCRIPTION:
Patients with psychotic disorders frequently require treatment at inpatient hospital settings during periods of acute illness for crisis management and stabilization. Although these patients often receive efficacious pharmacotherapy, there is a recognized lack of empirically-supported psychosocial interventions provided to patients in typical hospital settings. The provision of high quality psychosocial treatment during hospitalization is challenging due to short lengths of stay and a general lack of trained therapist employed on hospital units who can provide these evidence-based therapies. This unmet need for hospital psychosocial treatment represents a crucial missed opportunity to teach patients coping strategies that can speed time to recovery and impact post-discharge risk factors. Acceptance and Commitment Therapy (ACT) is a newer cognitive-behavioral approach that combines innovative mindfulness-based strategies for helping patients to cope more successfully with psychotic and other symptoms and implement values-consistent behavioral goals. However, adaptations to the original ACT approach are urgently needed to foster widespread implementation in community settings. The aim of the current study is to adapt the only promising acute-care psychosocial treatment for psychosis to be implementable in an inpatient setting and pilot test its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. current psychiatric hospitalization
2. diagnosis of schizophrenia, schizoaffective disorder, schizophreniform, brief psychotic disorder, delusional disorder, specified/unspecified other psychotic disorder, or a diagnosis of a mood disorder (major depressive disorder or bipolar disorder) with psychotic features, as determined by chart review and confirmed by the Structured Clinical Interview for Diagnostic and Statistical Manual (DSM)-5
3. 18 years or older
4. ability to speak and read English.

Exclusion Criteria:

1. psychosis severe enough to prevent participation in regular hospital groups
2. psychotic disorder related to a general medical condition or substance-induced psychotic disorder
3. significant cognitive impairment (mini-mental state exam score < 15).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-03; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale | Hospital Discharge (1 Week)

SECONDARY OUTCOMES:
Psychiatric Rehospitalization | 4 Months Post-Discharge

OTHER OUTCOMES:
Acceptance and Action Questionnaire-II | Hospital Discharge (1 Week)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Gaudiano, Ph.D., Principal Investigator — Butler Hospital/Brown University
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Gaudiano BA, Herbert JD. Acute treatment of inpatients with psychotic symptoms using Acceptance and Commitment Therapy: pilot results. Behav Res Ther. 2006 Mar;44(3):415-37. doi: 10.1016/j.brat.2005.02.007. PMID 15893293
- [Derived] Gaudiano BA, Ellenberg S, Johnson JE, Mueser KT, Miller IW. Effectiveness of acceptance and commitment therapy for inpatients with psychosis: Implementation feasibility and acceptability from a pilot randomized controlled trial. Schizophr Res. 2023 Nov;261:72-79. doi: 10.1016/j.schres.2023.09.017. Epub 2023 Sep 14. PMID 37716204